CLINICAL TRIAL: NCT05702242
Title: A Randomized Controlled Trial of No Strings Intrauterine Device (IUD) Removal Techniques: Alligator Forceps Versus Manual Vacuum Aspiration (MVA)
Brief Title: A Randomized Controlled Trial of No Strings Intrauterine Device (IUD) Removal Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2177
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: IUD Threads Not Visible; IUD Removal Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removal with alligator forceps (Experimental): Standard of care removal with passage of an intrauterine alligator forceps under ultrasound guidance to grasp and remove the IUD. If required, multiple attempts will be performed using this technique.
  Interventions: Procedure: IUD removal with no visible strings; Device: Alligator forceps
- Removal with manual vacuum aspiration (Experimental): Intrauterine placement of an MVA under ultrasound guidance adjacent to the IUD to remove the IUD. Multiple attempts will be performed up to a maximum of 3 unsuccessful MVA attempts, after which time, the provider will switch to the alligator forceps technique, given that this is the current standard of care.
  Interventions: Procedure: IUD removal with no visible strings; Device: Manual Vacuum Aspirator

INTERVENTIONS:
Procedure: IUD removal with no visible strings — Removal with either alligator forceps or MVA
Device: Alligator forceps — IUD removal with alligator forceps
  Arms: Removal with alligator forceps
Device: Manual Vacuum Aspirator — IUD removal with MVA
  Other Names: Ipas 60-mL double valve aspirator
  Arms: Removal with manual vacuum aspiration

SUMMARY:
The goal of this clinical trial is to compare success rates of two removal techniques for intrauterine devices (IUDs) that have missing or non-visible strings. The investigators will also collect preliminary data to better understand patient and provider satisfaction, maximum pain score, procedure time, and complications with the two techniques. Participants will be randomized to IUD removal with either an alligator forceps or manual vacuum aspiration (MVA) technique. This study will provide important data on these removal techniques, which could possibly expand options for and access to no strings IUD removals.

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are a commonly used, highly effective form of long-acting reversible contraception in the United States. Approximately 4-18% of people with an IUD in place with have missing or non-visible IUD strings, mostly commonly due to IUD string retraction into the cervix. Currently, expert opinion suggests to remove IUDs with no visible strings using by using an alligator forceps that is placed into the uterine cavity with or without ultrasound guidance. Removal of no strings IUDs with manual vacuum aspiration (MVA) has been suggested as a possible alternative to alligator forceps. MVA is a commonly used technique for the management of miscarriage, abortion, and endometrial sampling and has potential benefits as a low cost, portable device that is readily available in family planning clinic and many office-based obstetrics and gynecology practices.

The study will compare MVA to alligator forceps for IUD removal with no visible strings. The investigators will enroll females presenting for no strings IUD removals. Potential participants will be screened for eligibility and will be excluded if they have visible IUD strings, have a positive pregnancy test, have a partially retained IUD (e.g., IUD arm only), or are unwilling to be randomized to either arm. The investigators will perform a screening pelvic exam and transvaginal ultrasound (if not already completed prior to the visit). Participants will then be randomized to one of the two removal techniques: MVA or alligator forceps. The investigators will document successful removal with the first pass of the instrument as well as successful removal with multiple attempts of the same technique. A maximum of 3 MVA removal attempts will be performed after which time, the provider will switch to using an alligator forceps as the current standard of care. Preliminary data will also be collected on patient and provider satisfaction, patient pain scores, procedure time, and complications.

This study will provide important data on MVA as a technique for IUD removals with no visible strings. No studies have compared IUD removal techniques and expanding options for removal techniques has the potential to increase access to care.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18 - 45 years old
* Confirmed intrauterine IUD by pelvic ultrasound
* Desires IUD removal

Exclusion Criteria:

* Currently pregnant
* IUD strings are visible
* Partial retained IUD (e.g. IUD arm only)
* Unwilling to be randomized to either arm

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
First-pass IUD removal rates | 12-18 months
  To compare the first-pass intrauterine device (IUD) removal rates of using manual vacuum aspiration versus alligator forceps for IUD removal with no visible strings.

SECONDARY OUTCOMES:
Overall IUD removal success rates | 12-18 months
  To describe the overall success rates of IUD removal with no visible strings using alligator forceps versus manual vacuum aspiration.

OTHER OUTCOMES:
Preliminary data on satisfaction | 12-18 months
  To gather preliminary data on patient and provider satisfaction.
Preliminary data on pain scores | 12-18 months
  To gather preliminary data on maximum procedural pain scores measured by visual analog scale (VAS).
Preliminary data on procedure time | 12-18 months
  To gather preliminary data on total procedure time.
Preliminary data on complications | 12-18 months
  To gather preliminary data on complications of no strings IUD removals.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Clure, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Comprehensive Women's Health Center, Denver, Colorado, United States

REFERENCES:
- [Background] Prabhakaran S, Chuang A. In-office retrieval of intrauterine contraceptive devices with missing strings. Contraception. 2011 Feb;83(2):102-6. doi: 10.1016/j.contraception.2010.07.004. Epub 2010 Aug 23. No abstract available. PMID 21237334
- [Background] Marchi NM, Castro S, Hidalgo MM, Hidalgo C, Monteiro-Dantas C, Villarroeal M, Bahamondes L. Management of missing strings in users of intrauterine contraceptives. Contraception. 2012 Oct;86(4):354-8. doi: 10.1016/j.contraception.2012.01.018. Epub 2012 Mar 27. PMID 22459233
- [Background] Verma U, Astudillo-Davalos FE, Gerkowicz SA. Safe and cost-effective ultrasound guided removal of retained intrauterine device: our experience. Contraception. 2015 Jul;92(1):77-80. doi: 10.1016/j.contraception.2015.02.008. Epub 2015 Feb 21. PMID 25708503
- [Background] Swenson C, Royer PA, Turok DK, Jacobson JC, Amaral G, Sanders JN. Removal of the LNG IUD when strings are not visible: a case series. Contraception. 2014 Sep;90(3):288-90. doi: 10.1016/j.contraception.2014.04.007. Epub 2014 Apr 21. PMID 24835830
- [Background] Mizia K, Ramsay P. The effectiveness and safety of ultrasound-guided removal of a Mirena((R)) intrauterine system when the strings are not visible and conventional office procedures have failed. Aust N Z J Obstet Gynaecol. 2013 Aug;53(4):386-8. doi: 10.1111/ajo.12103. Epub 2013 Jun 26. PMID 23802598
- [Background] da Silva Nobrega AB, Pitangui ACR, Vieira CS. Factors associated with missing strings and expulsion after postplacental insertion of copper T380A intrauterine devices. Int J Gynaecol Obstet. 2022 Apr;157(1):67-75. doi: 10.1002/ijgo.13806. Epub 2021 Jul 27. PMID 34197636
- [Background] Wu JP, Porch E, Womack JP. Successful retrieval of an intrauterine device with "missing strings" using a manual vacuum aspirator in a desired early pregnancy: case report. J Minim Invasive Gynecol. 2011 Mar-Apr;18(2):254-6. doi: 10.1016/j.jmig.2010.11.008. PMID 21354074
- [Background] Jain A, Singh S, Elliyas S. Effectiveness of Manual Vacuum Aspiration (MVA) Device in the Management of Intrauterine Copper Devices (IUCD) with Missing Strings: A Prospective Interventional Study. J Obstet Gynaecol India. 2021 Aug;71(4):424-429. doi: 10.1007/s13224-021-01440-x. Epub 2021 Mar 15. PMID 34566303
- [Background] Guillebaud J, Kasonde JM. A simple scheme for managing the problem of 'lost threads' with intrauterine devices. Fertil Contracept. 1979 Apr;3(2):24-32. PMID 12309485